CLINICAL TRIAL: NCT06001229
Title: The Micheli Functional Scale's Validity and Reliability in Turkish Sport Groups
Brief Title: The Micheli Functional Scale's Validity and Reliability
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Aynur Demirel, Associate Professor, Hacettepe University
Other Study IDs: GO 22/540
Record Dates: First submitted 2023-08-14; First posted 2023-08-21 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to assess the reliability and validity of the "Micheli Functional Scale" in the Turkish context.

DETAILED DESCRIPTION:
The study will include a minimum of 80 individuals who are 16 years old or above, have been engaged in the same sports activity for at least two years, participate in physically demanding activities for at least three days a week, and possess the ability to read and write Turkish. Before participating in the study, athletes will be required to sign an informed consent form. Their demographic information will then be recorded.Before conducting the test, we will gather information about the athletes' history of low back pain using the extended Nordic musculoskeletal questionnaire. We will also use this questionnaire to identify any other musculoskeletal issues that the person may have.Two Turkish translators, fluent in English, will independently translate the original Micheli Functional Scale into Turkish. They will then discuss their translations and create a common one. The resulting translation will be translated back into English by two native English speakers who are also proficient in Turkish. These translations will be reviewed and combined into a single version. A Turkish scientist will evaluate the questionnaire for its suitability in the Turkish language. The final version will be tested on a small pilot group to determine its comprehensibility. After this, the questionnaire will be administered to the entire study group. To assess the validity of the Micheli Functional Scale, we will use the Oswestry Functional Questionnaire and the Ronald Morris Disability Questionnaire. One week after the test, we will repeat these surveys.

ELIGIBILITY:
Inclusion Criteria:

* 16 years old and over
* Having been doing the same sport for at least 2 years,
* Participating in sports activities or activities that require a high level of effort at least 3 days a week,
* Able to read and write Turkish

Exclusion Criteria:

* Has a cognitive problem that prevents him from understanding and answering the questions or is taking a drug that may cause them,
* Having a history of orthopedic or neurological injury or pain at a level that may prevent training or competition during the evaluation,
* History of spine/lower and upper extremity surgery,
* Structural deformities such as scoliosis and kyphosis,
* Those with trap neuropathy will be excluded from the study.

Ages: 16 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: To be eligible for the study, participants must be at least 16 years old, have been practicing the same sport for a minimum of 2 years, and engage in high-effort physical activity for at least 3 days per week. Additionally, those who are able to read and write in Turkish will be included in the study.
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2023-08-18 (Estimated); Primary Completion 2024-06-22 (Estimated); Study Completion 2024-06-22 (Estimated)

PRIMARY OUTCOMES:
Micheli Functional Scale | baseline and 1 week later
  Evaluates the function linked to low back pain in athletes.
Oswestry Disability Index | baseline and 1 week later
  Evaluate disability due to low back pain. the index measures perceived low back pain related dysfunction. Whether the total score increaeses, the dyscfunction increases.
Roland morris disability questionnaire | baseline and 1 week later
  It is a questionnaire used to evaluate the disability level of individuals with low back pain. This questionnaire, consisting of 24 items, questions the person's social life, walking, sitting, standing, getting up from a chair, climbing stairs, dressing, personal care, pain, appetite, sleep, and psychological impact. The person answers the questions with yes and no. Yes is scored as 1 point and no as 0 points. The maximum score is "24" and the minimum score is "0". As the total score increases, the level of physical exposure also increases.

SECONDARY OUTCOMES:
The musculoskeletal system problem | baseline
  Nordic Musculoskeletal System Questionnaire